CLINICAL TRIAL: NCT05552716
Title: Nationwide Study of Firearm Violence Prevention Tactics and Policies in K-12 Schools
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Charles Branas, Gelman Professor of Epidemiology, Chair, Department of Epidemiology, Columbia University
Other Study IDs: AAAT9087; 1R01HD108027-01 (NIH)
Record Dates: First submitted 2022-09-21; First posted 2022-09-23 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Violence
Keywords: Gun violence; Child health; School safety; Firearm violence prevention tactics and policies
MeSH Terms: interventions — Policy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case Schools: All Schools identified with all incidents in which a gun is fired, or a bullet hits school property for any reason, regardless of the number of victims, time, day of the week.
  Interventions: Other: School safety tactics and policies
- Control Schools: A random sample of schools that have not experienced any incidents in which a gun is fired, or a bullet hits school property for any reason, regardless of the number of victims, time, day of the week matched with a case school based on geographic state, urban/non-urban status, and elementary/middle/high school status.
  Interventions: Other: School safety tactics and policies

INTERVENTIONS:
Other: School safety tactics and policies — A list of school safety tactics and policies (such as metal detectors, armed security guards, active shooter drills) that were in place at the school at the time of shooting.

SUMMARY:
This observational study will collect data and address the following three specific aims.

Aim 1: To determine if the total number and specific types of safety tactics and policies are associated with the occurrence of intentional shootings in a sample of 650+ K-12 public schools.

Primary Aim 1 hypothesis -- The total number of cumulative safety tactics and policies will be significantly associated with intentional school shootings.

Secondary Aim 1 hypothesis -- When organized into three domains (physical target hardening, emergency response and technologies, and school security), the total number of safety tactics and policies within each domain will be significantly associated with intentional school shootings.

Aim 2: To determine if the total number and specific types of safety tactics and policies are associated with suspension and expulsion rates in a sample of 650+ K-12 public schools.

Primary Aim 2 hypothesis -- The total number of cumulative safety tactics and policies will be significantly associated with student discipline outcomes.

Secondary Aim 2 hypothesis -- When organized into three domains (physical target hardening, emergency response and technologies, and school security), the total number of safety tactics and policies within each domain will be significantly associated with student discipline outcomes.

Aim 3: To identify if urban/non-urban, economic, and racial disparities prior to and following the onset of the COVID-19 pandemic exist in effect modification analyses of the relationships between the implementation of safety tactics and policies, suspensions and expulsions, and intentional shootings in K-12 public schools.

Aim 3 Hypothesis: Significant urban/non-urban, economic, and racial disparities prior to and following the onset of the COVID-19 pandemic will exist in effect modification analyses of the relationships between the implementation of safety tactics and policies, suspensions and expulsions, and intentional shootings in K-12 public schools.

DETAILED DESCRIPTION:
Firearm violence in K-12 schools is a persistent public health threat in the US. The negative impact of these tragedies on children and school staff is significant. School-wide efforts (e.g. metal detectors, active shooter drills, armed school personnel, and two dozen others) to improve safety and assuage fears are being widely implemented in public K-12 schools across the US. Yet, the effectiveness of most of these strategies at deterring school shootings has never been scientifically tested. Moreover, school districts may differentially use these strategies based on factors unrelated to school safety, including as a means to discipline students. These gaps in evidence are particularly significant, as the U.S. K-12 public school system currently serves an estimated 51 million children. The proposed research team has conducted pilot and preliminary research demonstrating the feasibility of the larger study proposed here.

This will be accomplished through a nationally representative, population-based, case-control study comparing hundreds of case schools that have experienced a school shooting and randomly selected control schools that have not experienced such an event using epidemiological incidence density sampling. Case data will be ascertained primarily via the FEMA-funded Naval Postgraduate School K-12 School Shooting database. Additional databases that record and publicly report school shooting incidents will be linked and harmonized. One control school will be randomly selected from a national database of public K-12 schools at the National Center for Education Statistics and matched to each case school based on state, urban/nonurban, and elementary/middle/high school status. Both case and control schools will have a list of school safety tactics and policies that were in place, or not in the case school at the time of shooting and the control schools during same time period.

Publicly accessible school safety plans and multiple publicly available secondary sources of data will be used to determine the safety strategies in place at both case and control schools during the school year before each case school's shooting event. These data will be linked to data on school suspensions and expulsions, obtained from the national Civil Rights Data Collection effort. Results will newly inform school policies and practices to reduce gun violence and promote healthy experiences for children across disparate school communities.

ELIGIBILITY:
For a case school to be included, it must satisfy the following criteria:

Inclusion Criteria-

1. The incident must have taken place on the school property.
2. The gun must have been shot during school hours.

Exclusion Criteria:

1. The shot was accidental.
2. If it was a suicide/attempted suicide and there was no attempt to shoot another person. (Murder-suicides will be included.)
3. The shot was fired on the school bus on its way to or from the school or another school-sanctioned event.
4. The school was not in session for any reason.
5. The school event was taking place at a location where school security measures were ineffective.
6. The shot originated from outside the school and no person or property was hit in the school.

Inclusion criteria for control school: Matches the case school on the following criteria- geographic state, urban/non-urban, and elementary/middle/high school status.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The large majority of data collected in this proposed study does not involve human subjects. Nearly all (if not all) data collected in this study will be publicly available. In the case that a school's safety plan for a specific academic year of interest is not available online, the MPIs will email the principal of the school directly to inquire if they would be willing to provide a copy of the safety plan for the purpose of this research study. As a result, the principal of every participating school in this proposed work will be eligible for participation.
Sampling Method: Probability Sample
Enrollment: 648 (Actual)
Dates: Start 2023-05-11 (Actual); Primary Completion 2025-01-20 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
Occurrence of School Shooting | Up to 9 years (January, 01, 2015 to December 31, 2023)
  School shooting is described as a gun being discharged on the school premises during the school hours.

SECONDARY OUTCOMES:
Occurrence of Student Discipline | Up to 9 years (January, 01, 2015 to December 31, 2023)
  Student discipline is defined as the number of suspensions, and number of expulsions.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Branas, PhD, Principal Investigator — Mailman School of Public Health
Locations (1):
- Columbia Mailman School of Public Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No